CLINICAL TRIAL: NCT06893926
Title: Evaluating the Utility of S100B Protein Concentration for Diagnosing Fetal Central Nervous System Hypoxia-Ischemia in Children With Late Fetal Growth Retardation: A Prospective Cohort Study
Brief Title: Cord Blood S100B Protein Concentration in Neonates With Fetal Growth Restriction
Status: Recruiting | Type: Observational
Sponsor: Institute of Mother and Child, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Agnieszka Drozdowska-Szymczak, MD, PhD, Institute of Mother and Child, Warsaw, Poland
Other Study IDs: S100BFGR
Record Dates: First submitted 2025-03-06; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: s100b; Hypoxia-Ischemia, Brain; Fetal Growth Restriction (FGR)
Keywords: S100B protein; fetal growth restriction (FGR); newborn; central nervous system (CNS) damage; CNS hypoxia-ischemia (HI)
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Women with a full-term pregnancy and a prenatal diagnosis of late-onset FGR.
  Interventions: Diagnostic Test: Prenatal ultrasound examination with blood flow analysis; Diagnostic Test: Umbilical cord blood gas analysis; Diagnostic Test: Umbilical cord blood S100B protein level; Diagnostic Test: Neonatal transfontanelle ultrasound assessment
- Control group: Women with a full-term pregnancy and normal fetal development.
  Interventions: Diagnostic Test: Prenatal ultrasound examination with blood flow analysis; Diagnostic Test: Umbilical cord blood gas analysis; Diagnostic Test: Umbilical cord blood S100B protein level; Diagnostic Test: Neonatal transfontanelle ultrasound assessment

INTERVENTIONS:
Diagnostic Test: Prenatal ultrasound examination with blood flow analysis — For all patients who provide informed consent to participate in the study, an ultrasound examination is performed within 48 hours prior to delivery. This assessment includes:
  1. Measurement of fetal anthropometric parameters and estimation of fetal weight.
  2. Evaluation of blood flow using the pulsatility index (PI) in the UA, UtA, DV, and MCA.
Diagnostic Test: Umbilical cord blood gas analysis — A 0.5 mL blood sample is collected from the clamped section of the umbilical cord and immediately sent to the laboratory for cord blood gas analysis, including the determination of pH, base excess (BE), and lactate levels.
Diagnostic Test: Umbilical cord blood S100B protein level — A 1 mL sample of cord blood is collected in a labeled tube, which includes the mother's name, the child's gender, date of birth, and date of collection. The sample is then sent to the laboratory for centrifugation. The resulting serum samples are frozen, and once approximately 80 samples have been collected, they will be thawed and analyzed for S100B protein concentration. Any remaining material after laboratory processing will be properly disposed of.
Diagnostic Test: Neonatal transfontanelle ultrasound assessment — A transfontanelle ultrasound examination is performed to assess for any abnormalities in the newborn.

SUMMARY:
S100B protein is a biomarker that increases following central nervous system (CNS) damage. Measuring this protein's levels may allow for the early identification of infants at high risk for developmental abnormalities, such as fetal growth restriction (FGR), even on the first day of life, in a non-invasive manner. Early detection could enable timely interventions and rehabilitation, potentially improving the child's prognosis and long-term outcomes. This study investigates two groups of full-term pregnancies: a study group with prenatally diagnosed late FGR, and a control group with normal fetal growth. Following delivery, cord blood samples from both groups will be analyzed for S100B protein concentrations, pH, base excess (BE), and lactate levels. Additionally, fetal blood flow parameters in the umbilical artery (UA), uterine arteries (UtA), ductus venosus (DV), and middle cerebral artery (MCA) will be monitored via ultrasound within 48 hours before delivery. This study aims to compare S100B protein concentrations in umbilical cord blood between the two groups and to assess correlations with fetal Doppler parameters, pH, BE, and lactate levels in cord blood gas analysis. Ultimately, we seek to determine the effectiveness of S100B protein concentration as a biomarker for diagnosing fetal CNS hypoxia- ischemia in FGR-affected children, compared to those with normal growth.

ELIGIBILITY:
Study Group - Inclusion Criteria:

1. Women with a full-term pregnancy (≥37 weeks of gestation), singleton.
2. Pregnancy complicated by FGR.

Study Group - Exclusion Criteria:

1. Antenatal (at recruitment):

   * Maternal conditions that may affect the blood flow in placental vessels, including smoking, use of illicit stimulant substances, or pregestational diabetes.
   * Maternal depression requiring pharmacological treatment (e.g., SSRIs).
2. Intrapartum:

   * Factors indicating a possible intrauterine infection, such as amniotic fluid leakage for more than 15 hours, spontaneous preterm labor, diagnosed intrauterine infection, or symptoms of infection in the mother.
   * Prolonged labor lasting more than 15 hours.

Control Group - Inclusion Criteria:

1. Women with a full-term pregnancy (≥37 weeks of gestation), singleton.
2. Pregnancy not complicated by FGR.

Control Group - Exclusion Criteria:

1. Antenatal (at recruitment):

   * Maternal conditions that may affect placental blood flow, such as smoking, use of illicit stimulant substances, pregestational diabetes, or chronic hypertension.
   * Maternal depression requiring pharmacological treatment (e.g., SSRIs).
   * Risk factors for intrauterine HI, including abnormal fetal blood flow parameters on ultrasound, abnormal CTG recordings, or the need for intrauterine transfusion.
2. Intrapartum:

   * Indicators of possible intrauterine infection, such as amniotic fluid leakage for more than 15 hours, spontaneous preterm delivery, diagnosed intrauterine infection, or maternal symptoms of infection.
   * Risk factors for perinatal HI.
   * Prolonged labor lasting more than 15 hours (counted from the onset of regular uterine contractions).
   * Birth weight below the 10th percentile or above the 90th percentile.
   * Apgar score less than 8 at the 1st, 3rd, 5th, or 10th minute of life.
   * Abnormal umbilical cord blood gas analysis results, defined as pH < 7.15 or BE < -9.3 mmol/l.
3. Postnatal:

   * Neonatal anemia requiring a top-up transfusion within the first 24 hours of life

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with a full-term pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Cord blood S100B protein concentration | Within 3 months of enrollment
  The study's primary endpoint will be the concentration of S100B protein measured from a cord blood sample taken after birth in both the study and control groups.

SECONDARY OUTCOMES:
Correlation of cord blood S100B concentration with pH, BE, and lactate levels in cord blood gas analysis | Within 3 months of enrollment
  The potential correlation between cord blood S100B concentration and pH, BE, and lactate levels, as determined by cord blood gas analysis, in both the study and control groups.
Association between cord blood S100B protein concentration and fetal blood flow parameters | Within 3 months of enrollment
  The potential relationship between cord blood S100B protein concentration and blood flow parameters (PI) in the UA, UtA, DV, and MCA, as assessed by fetal ultrasound performed within 48 hours before delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka A. Drozdowska-Szymczak, MD, PhD, Principal Investigator — Institute of Mother and Child in Warsaw, Poland
Locations (1):
- Institute of Mother and Child, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mazarico E, Llurba E, Cumplido R, Valls A, Melchor JC, Iglesias M, Cabero L, Gratacos E, Gomez-Roig MD. Neural injury markers in intrauterine growth restriction and their relation to perinatal outcomes. Pediatr Res. 2017 Sep;82(3):452-457. doi: 10.1038/pr.2017.108. Epub 2017 May 31. PMID 28426650
- [Background] Strzalko B, Karowicz-Bilinska A, Wyka K, Krajewski P, Kesiak M, Kociszewska-Najman B. Serum S100B Protein Concentrations in SGA/FGR newborns. Ginekol Pol. 2021 Jun 9. doi: 10.5603/GP.a2021.0119. Online ahead of print. PMID 34105746
- [Background] Malhotra A, Ditchfield M, Fahey MC, Castillo-Melendez M, Allison BJ, Polglase GR, Wallace EM, Hodges R, Jenkin G, Miller SL. Detection and assessment of brain injury in the growth-restricted fetus and neonate. Pediatr Res. 2017 Aug;82(2):184-193. doi: 10.1038/pr.2017.37. Epub 2017 May 17. PMID 28234891
- [Background] Zaigham M, Lundberg F, Olofsson P. Protein S100B in umbilical cord blood as a potential biomarker of hypoxic-ischemic encephalopathy in asphyxiated newborns. Early Hum Dev. 2017 Sep;112:48-53. doi: 10.1016/j.earlhumdev.2017.07.015. Epub 2017 Jul 27. PMID 28756088
- [Background] Bouvier D, Giguere Y, Pereira B, Bernard N, Marc I, Sapin V, Forest JC. Cord blood S100B: reference ranges and interest for early identification of newborns with brain injury. Clin Chem Lab Med. 2020 Jan 28;58(2):285-293. doi: 10.1515/cclm-2019-0737. PMID 31622243
- [Background] Velipasaoglu M, Yurdakok M, Ozyuncu O, Portakal O, Deren O. Neural injury markers to predict neonatal complications in intrauterine growth restriction. J Obstet Gynaecol. 2015;35(6):555-60. doi: 10.3109/01443615.2014.978848. Epub 2014 Nov 13. PMID 25392968
- [Background] Perrone S, Grassi F, Caporilli C, Boscarino G, Carbone G, Petrolini C, Gambini LM, Di Peri A, Moretti S, Buonocore G, Esposito SMR. Brain Damage in Preterm and Full-Term Neonates: Serum Biomarkers for the Early Diagnosis and Intervention. Antioxidants (Basel). 2023 Jan 29;12(2):309. doi: 10.3390/antiox12020309. PMID 36829868
- [Background] Chiang LM, Chen WY, Yang YC, Jeng MJ. Elevation of serum S100 protein concentration as a marker of ischemic brain damage in extremely preterm infants. J Chin Med Assoc. 2015 Oct;78(10):610-6. doi: 10.1016/j.jcma.2015.06.009. Epub 2015 Aug 15. PMID 26285828
- [Background] Florio P, Abella R, Marinoni E, Di Iorio R, Li Volti G, Galvano F, Pongiglione G, Frigiola A, Pinzauti S, Petraglia F, Gazzolo D. Biochemical markers of perinatal brain damage. Front Biosci (Schol Ed). 2010 Jan 1;2(1):47-72. doi: 10.2741/s45. PMID 20036928
- [Background] Huang RZ, Zhang YJ, Zhang JF, Su YM, Peng LQ, Ya N. Relation between prognosis and changes of MBP and S100B in premature infants with periventricular leukomalacia. Genet Mol Res. 2015 Apr 30;14(2):4338-43. doi: 10.4238/2015.April.30.6. PMID 25966206
- [Background] Metallinou D, Karampas G, Lazarou E, Iacovidou N, Pervanidou P, Lykeridou K, Mastorakos G, Rizos D. Serum Activin A as Brain Injury Biomarker in the First Three Days of Life. A Prospective Case-Control Longitudinal Study in Human Premature Neonates. Brain Sci. 2021 Sep 20;11(9):1243. doi: 10.3390/brainsci11091243. PMID 34573263
- [Background] Lu H, Huang W, Chen X, Wang Q, Zhang Q, Chang M. Relationship between premature brain injury and multiple biomarkers in cord blood and amniotic fluid. J Matern Fetal Neonatal Med. 2018 Nov;31(21):2898-2904. doi: 10.1080/14767058.2017.1359532. Epub 2017 Aug 3. PMID 28738706
- [Background] Friel LA, Romero R, Edwin S, Nien JK, Gomez R, Chaiworapongsa T, Kusanovic JP, Tolosa JE, Hassan SS, Espinoza J. The calcium binding protein, S100B, is increased in the amniotic fluid of women with intra-amniotic infection/inflammation and preterm labor with intact or ruptured membranes. J Perinat Med. 2007;35(5):385-93. doi: 10.1515/JPM.2007.101. PMID 17624933
- [Background] Niwa Y, Imai K, Kotani T, Miki R, Nakano T, Ushida T, Moriyama Y, Kikkawa F. Relationship between cytokine profiles of cord blood and cord S100B levels in preterm infants. Early Hum Dev. 2019 Feb;129:65-70. doi: 10.1016/j.earlhumdev.2019.01.013. Epub 2019 Jan 23. No abstract available. PMID 30684905
- [Background] Wirds JW, Duyn AE, Geraerts SD, Preijer E, Van Diemen-Steenvoorde JA, Van Leeuwen JH, Haas FJ, Gerritsen WB, De Boer A, Leusink JA. S100 protein content of umbilical cord blood in healthy newborns in relation to mode of delivery. Arch Dis Child Fetal Neonatal Ed. 2003 Jan;88(1):F67-9. doi: 10.1136/fn.88.1.f67. PMID 12496231
- [Background] Masaoka N, Nakajima Y, Morooka M, Tashiro H, Wada M, Maruta K, Iwane E, Yamashiro M. The impact of intrauterine infection on fetal brain damage assessed by S100B protein concentrations in umbilical cord arteries. J Matern Fetal Neonatal Med. 2016;29(15):2464-9. doi: 10.3109/14767058.2015.1087501. Epub 2015 Sep 30. PMID 26421445
- [Background] Schulpis KH, Margeli A, Akalestos A, Vlachos GD, Partsinevelos GA, Papastamataki M, Antsaklis A, Papassotiriou I. Effects of mode of delivery on maternal-neonatal plasma antioxidant status and on protein S100B serum concentrations. Scand J Clin Lab Invest. 2006;66(8):733-42. doi: 10.1080/00365510600977737. PMID 17101566
- [Background] Pawluski JL, Galea LA, Brain U, Papsdorf M, Oberlander TF. Neonatal S100B protein levels after prenatal exposure to selective serotonin reuptake inhibitors. Pediatrics. 2009 Oct;124(4):e662-70. doi: 10.1542/peds.2009-0442. Epub 2009 Sep 28. PMID 19786426
- [Background] Eixarch E, Meler E, Iraola A, Illa M, Crispi F, Hernandez-Andrade E, Gratacos E, Figueras F. Neurodevelopmental outcome in 2-year-old infants who were small-for-gestational age term fetuses with cerebral blood flow redistribution. Ultrasound Obstet Gynecol. 2008 Dec;32(7):894-9. doi: 10.1002/uog.6249. PMID 19035538
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. J Clin Epidemiol. 2008 Apr;61(4):344-9. doi: 10.1016/j.jclinepi.2007.11.008. PMID 18313558
- [Background] Cuschieri S. The STROBE guidelines. Saudi J Anaesth. 2019 Apr;13(Suppl 1):S31-S34. doi: 10.4103/sja.SJA_543_18. PMID 30930717
- [Background] Fenton TR, Kim JH. A systematic review and meta-analysis to revise the Fenton growth chart for preterm infants. BMC Pediatr. 2013 Apr 20;13:59. doi: 10.1186/1471-2431-13-59. PMID 23601190
- [Background] Kwiatkowski S, Torbe A, Borowski D, Breborowicz G, Czajkowski K, Huras H, Kajdy A, Kalinka J, Kosinska-Kaczynska K, Leszczynska-Gorzelak B, Rokita W, Ropacka-Lesiak M, Sieroszewski P, Wielgos M, Zimmer M. Polish Society of Gynecologists and Obstetricians Recommendations on diagnosis and management of fetal growth restriction. Ginekol Pol. 2020;91(10):634-643. doi: 10.5603/GP.2020.0158. No abstract available. PMID 33184833
- [Background] Gordijn SJ, Beune IM, Thilaganathan B, Papageorghiou A, Baschat AA, Baker PN, Silver RM, Wynia K, Ganzevoort W. Consensus definition of fetal growth restriction: a Delphi procedure. Ultrasound Obstet Gynecol. 2016 Sep;48(3):333-9. doi: 10.1002/uog.15884. PMID 26909664
- [Background] Gazzolo D, Abella R, Marinoni E, di Iorio R, Li Volti G, Galvano F, Frigiola A, Temporini F, Moresco L, Colivicchi M, Sabatini M, Ricotti A, Strozzi MC, Crivelli S, Risso FM, Sannia A, Florio P. New markers of neonatal neurology. J Matern Fetal Neonatal Med. 2009;22 Suppl 3:57-61. doi: 10.1080/14767050903181468. PMID 19718579